CLINICAL TRIAL: NCT07257003
Title: A Nationwide Multicenter, Single-arm, Retrospective Study on Delayed Endoscopic Direct-to-implant Breast Reconstruction Via Axillary Approach After Simple Mastectomy in Breast Cancer Patients
Brief Title: A Nationwide Multicenter, Single-arm, Retrospective Study of Delayed Endoscopic DTI-BR After Simple Mastectomy
Acronym: DEDTI-BR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Du Zhenggui (Other)
Collaborators: Fujian Cancer Hospital (Other Government); Suzhou Municipal Hospital (Other); The Second People's Hospital of Yibin (Other); Mianyang Central Hospital (Other); West China Fourth Hospital, Sichuan University (Unknown); The Fourth People's Hospital of Sichuan Province (Unknown)
Responsible Party: Sponsor-Investigator, Du Zhenggui, Deputy director. Zhenggui Du, West China Hospital
Organization: West China Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025(1896)
Record Dates: First submitted 2025-11-14; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Endoscopic surgery; Breast reconstruction; Minimal invasive surgery
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DEDTI-BR group (Experimental): delayed endoscopic direct-to-implant breast reconstruction via axillary approach after simple mastectomy
  Interventions: Procedure: delayed endoscopic direct-to-implant breast reconstruction via axillary approach after simple mastectomy

INTERVENTIONS:
Procedure: delayed endoscopic direct-to-implant breast reconstruction via axillary approach after simple mastectomy — This technique allows for breast reconstruction in a single operation. Taking dual-plane breast reconstruction as an example, preoperative marking lines are drawn to indicate the contour and inframammary fold of the reconstructed breast. A 4-5 cm axillary incision is placed one finger-breadth below the axillary apex. After making the skin incision, the plane between the pectoralis major and minor muscles is identified and dissected, extending approximately 2 cm below the previous mastectomy horizontal scar. The inner and lower parts of the pectoralis major muscle were then separated. Proceed to the subcutaneous layer and continue to dissociate the flap until it reaches the pre-designed folds and the breast boundary. The use of the TiLOOP® Bra depends on the thickness of the patient's flap. Finally, the prosthesis is placed behind the pectoralis major muscle for breast reconstruction.

SUMMARY:
This study is a nationwide multicenter, single-arm, retrospective study. The study aims to conduct a detailed analysis of operation-related parameters, aesthetic outcomes (e.g., BREAST-Q scores and Harris scores), and safety (e.g., surgical complication rates) in delayed endoscopic direct-to-implant breast reconstruction via the axillary approach.

DETAILED DESCRIPTION:
Breast cancer is the most common malignancy in women, with mastectomy remaining the predominant surgical approach in many regions-often leaving patients with psychological distress from breast loss. With the progress of treatment, patients' survival is prolonged and their quality of life is improved, so the demand for breast reconstruction is increasing. The two-stage implant-based breast reconstruction (TS-IBR) often needs two procedures, two anesthetics, and multiple hospital visits for the injection of water into the expander-costs that increase both financially and in time, ultimately affecting their work and daily routines. Ultimately, whether the procedure reopens the original scar or makes a new incision on the chest-and despite the skin being gradually expanded using an expander-there remains a high risk of dehiscence, implant exposure, infection, and even implant removal. Another method for breast reconstruction after total mastectomy is autologous breast reconstruction (ABR), which doesn't need a second operation. Still, it has serious scar problems and increases the risk of donor-site trauma and complications. Additionally, sensation and function at the donor site may be somewhat reduced, and both sites will likely have large scars, which can significantly impact the aesthetic results.

Therefore, the investigators need to find a simple, efficient, and safe method. The investigators developed the reverse-sequence endoscopic nipple-sparing mastectomy (R-E-NSM) with direct-to-implant breast reconstruction (DIBR), which changes the surgical sequence, makes the operation simple, and realizes immediate breast reconstruction. Inspired by endoscopic breast augmentation methods through the axillary incision, our team also developed a novel technique called delayed endoscopic direct-to-implant breast reconstruction (DEDTI-BR). Clinical practice shows that this technique is also suitable for patients after total mastectomy. This technique utilizes seroma for natural skin expansion, eliminates secondary operations, and preserves aesthetics without additional scars-significantly improving patients' quality of life. Despite its theoretical benefits, clinical evidence validating its efficacy and safety is currently lacking.

Therefore, the investigators plan to conduct a nationwide, multicenter, single-arm, retrospective study, analyzing operation-related parameters, aesthetic outcomes (e.g., BREAST-Q scores and Harris scores), and safety (e.g., surgical complication rates) in DEDTI-BR via the axillary approach. Our goal is to inform and guide clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients who underwent delayed endoscopic direct-to-implant breast reconstruction after simple mastectomy at various centers from July 2024 to August 2025, all delayed endoscopic direct-to-implant breast reconstructions were performed ≥ 6 months after the initial mastectomy.

Exclusion Criteria:

* Poor skin elasticity;
* Re-evaluation (based on clinical, imaging, and pathological findings) indicates local or regional recurrence or uncontrolled distant metastasis;
* Patients who have previously undergone radical mastectomy;
* Patients who refused to provide postoperative follow-up information.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The patient's satisfaction with the breasts | postoperative 6-month
  Satisfaction with the breast of the BREAST-Q scale. The BREAST-Q is commonly used to assess health-related satisfaction and quality of life in patients who have undergone breast reconstruction after mastectomy. Responses for each subscale are scored from 0 to 100, with higher scores indicating better outcomes.

SECONDARY OUTCOMES:
The surgical safety | postoperative 6-month
  Surgical complication rates, including flap scald, NAC ischemia/necrosis, seroma, surgical area infection, bleeding, incision splitting, flap ischemia/necrosis
The aesthetic outcomes | postoperative 6-month
  BREAST-Q scale (physical well-being: chest, psychosocial well-being, sexual well-being) and Harris scale. The BREAST-Q is commonly used to assess health-related satisfaction and quality of life in patients who have undergone breast reconstruction after mastectomy. Responses for each subscale are scored from 0 to 100, with higher scores indicating better outcomes. The Harris score is used to evaluate the postoperative cosmetic outcome, which is classified as excellent, good, general, and poor.
The implant-assisted complications | postoperative 6-month
  Implant-assisted complication rates, including rippling, prosthesis outline appearance, capsular contraction, animation deformity, pectoralis major pain, pectoralis major muscle spasm

CONTACTS AND LOCATIONS:
Locations (1):
- West China hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data via the request portal. All IPD requests should be emailed to Dr. Zhenggui Du, the general project leader, and will be evaluated by Dr. Du and the head of the collaborating organization to decide whether to approve.
Supporting Information: Study Protocol, SAP
Time Frame: After publication of relevant research outputs, such as academic papers and books.
Access Criteria: When a request has been approved, the investigator will provide access to the de-identified individual patient-level data in the data management platform (Electronic Data Capture, EDC). A signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing the requested information. Additionally, all users will need to accept the terms and conditions of the data management platform to gain access.
URL: https://dct.meddb.cn/login_index

REFERENCES:
- [Background] Xiu B, Zhang Q, Meng X, Hao S, Yang B, Li J, Shao ZM, Wu J; Chinese Anti-Cancer Association; Committee of Breast Cancer Society. Current practices and challenges of endoscopic-assisted breast surgery in China: A nationwide cross-sectional survey. Eur J Surg Oncol. 2025 May;51(5):109620. doi: 10.1016/j.ejso.2025.109620. Epub 2025 Jan 19. PMID 39842261
- [Background] Bennett KG, Qi J, Kim HM, Hamill JB, Pusic AL, Wilkins EG. Comparison of 2-Year Complication Rates Among Common Techniques for Postmastectomy Breast Reconstruction. JAMA Surg. 2018 Oct 1;153(10):901-908. doi: 10.1001/jamasurg.2018.1687. PMID 29926077
- [Background] Ren Y, Yu Y, Xu K, Li Z, Wang X. Meta-Analysis of Immediate Implant-Based Breast Reconstruction Versus Autologous Breast Reconstruction in the Setting of PMRT. Aesthetic Plast Surg. 2024 May;48(10):1940-1948. doi: 10.1007/s00266-023-03430-y. Epub 2023 Jun 28. PMID 37380747
- [Background] Movassaghi K, Gilson A, Stewart CN, Cusic J, Movassaghi A. Prepectoral Two-Stage Implant-Based Breast Reconstruction with Poly-4-Hydroxybutyrate for Pocket Control without the Use of Acellular Dermal Matrix: A 4-Year Review. Plast Reconstr Surg. 2024 Jul 1;154(1):15-24. doi: 10.1097/PRS.0000000000010914. Epub 2023 Jul 6. PMID 37410610
- [Background] Deliere A, Attai D, Victorson D, Kuchta K, Pesce C, Kopkash K, Sisco M, Seth A, Yao K. Patients Undergoing Bilateral Mastectomy and Breast-Conserving Surgery Have the Lowest Levels of Regret: The WhySurg Study. Ann Surg Oncol. 2021 Oct;28(10):5686-5697. doi: 10.1245/s10434-021-10452-w. Epub 2021 Aug 25. PMID 34432189
- [Background] Erden Y, Celik HC, Karakurt N. Women's body image after mastectomy: a photovoice study. Support Care Cancer. 2025 May 27;33(6):501. doi: 10.1007/s00520-025-09541-3. PMID 40423833